CLINICAL TRIAL: NCT06051539
Title: Outcomes and Health Economics of Stroke Using Rhythmic Auditory Stimulation
Acronym: OrcHESTRAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedRhythms, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PS300
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Intervention Model Description: The study will follow a withdrawal with randomized re-treatment design. The study will consist of two steps. In Step 1, all participants will receive the MR-001 intervention for 12 weeks, followed by a 12-week washout period. At Step 2, participants will be randomized to receive either another 12 weeks of intervention followed by another 12-week washout or continue their first washout for an additional 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort A: Restart Intervention (Experimental): Participants in Cohort A will perform active walking for 30 minutes at a time with MR-001, at least 3 times a week, for 12 weeks in their home/community environment.
  Interventions: Device: MR-001
- Cohort B: Continued Washout (No Intervention): Participants in Cohort B will continue their washout period for another 24 weeks.

INTERVENTIONS:
Device: MR-001 — MR-001 is an autonomous neurorehabilitation system based on the principles of Rhythmic Auditory Stimulation intended to improve walking and ambulation in adult chronic stroke patients. MR-001 is intended to be a prescription use only device for use at home/community. The user operates the MR-001 System autonomously and the therapy progresses automatically once a user engages in a session. The MR-001 system consists of two foot sensors that measure walking, a touchscreen device preloaded solely with a proprietary software application, a headset, and charging equipment. The electronic components are powered by lithium-ion rechargeable batteries. Participants are asked to walk with the device for 3 times per week for 12 weeks. Each walking session is 30 minutes in length.
  Arms: Cohort A: Restart Intervention

SUMMARY:
The purpose of this trial is to assess engagement, efficacy, durability, and impact on health care resource utilization of MR-001 in persons with chronic stroke who have a gait deficit after in-home/community use.

DETAILED DESCRIPTION:
This is a decentralized clinical trial designed to assess clinical outcomes and resulting healthcare resource utilization (HCRU) of MedRhythms' MR-001 device used by patients with chronic stroke in the home setting.

MR-001 is an autonomous neurorehabilitation system based on the principles of Rhythmic Auditory Stimulation intended to improve walking in adult chronic stroke patients. MR-001 is a prescription medical device intended for use at home. The user operates the device autonomously and the therapy progresses automatically once a user engages in a session.

The MR-001 system consists of two foot sensors that measure walking, a locked touchscreen device preloaded with a proprietary software application, a headset, and charging equipment. The electronic components are powered by lithium-ion rechargeable batteries.

The primary objective of this study is to assess engagement with MR-001 walking therapy in chronic stroke patients with a gait deficit in a real world setting. The primary endpoint will be measured by session completion over the 12 week intervention period. Secondary endpoints include assessing effect on walking endurance, durability of response, and reintroduction of the intervention, as well as effect on healthcare resource utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Equal to or greater than 6 months post-stroke with gait impairment
2. Age >/= 18 - 85 years of age, inclusive
3. Understand and speak English
4. Must be able to ambulate without assistance from another person. Note: assistive devices are allowed. If a participant uses an assistive device at the time of enrollment, the device must be used for all walking sessions.
5. Willing to travel to a Velocity location to complete in-person gait assessments
6. Able to walk at a speed greater than or equal to 0.4 m/s as derived as an average of speed per minute from the 6MWT. Note: if a participant intends to use an assistive device throughout the intervention period, the assistive device must be used during the gait assessment.
7. Must have claims data available and consent to sharing.

Exclusion Criteria:

1. Hearing impairment with or without the use of hearing aids such that the participant cannot hear the rhythmic stimulation of the music
2. Pain that impairs walking ability
3. Unable to safely participate in walking sessions as determined by investigator
4. Requires more than one rest (seated or not) during the 6MWT
5. Significant comorbid medical or neurological conditions that could impact gait or prevent safe participation as determined by the Investigator. For example: condition that prevents participation in exercise, e.g., Parkinson's disease, cerebral palsy, multiple sclerosis, myasthenia gravis, muscular dystrophy, or spinal cord injury. Note: major surgery within the last 3 months is exclusionary.
6. People who are pregnant or become pregnant (due to expected gait pattern changes).
7. Lower limb prosthetic
8. More than 2 falls in the previous month
9. Non-reciprocal gait pattern. Note: Note: a non-reciprocal gait pattern is defined as a 3-point step pattern. Participants must have a 2-point step pattern to qualify. Asymmetry seen in gait is acceptable.
10. Treatment with a gait-based investigational intervention within the last 3 months.
11. Unable or unwilling to provide informed consent to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of walking sessions during 12-week intervention period | 12 weeks
  The purpose of this study is to assess engagement with MR-001 walking therapy in chronic stroke patients with a gait deficit in a real world setting. Engagement will be measured as number of walking sessions observed across the 12 week intervention period.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | From baseline to end of treatment at 12 weeks
  To assess whether MR-001 improves walking endurance after 12 weeks of treatment
6 Minute Walk Test (6MWT) | At 16 and 24 weeks
  To assess durability of walking endurance response to MR-001 after 12 weeks of intervention
Patient Health Questionnaire-8 (PHQ-8) | 12 weeks
  To assess whether MR-001 improves health-related quality of life in chronic stroke patients with gait deficit
The Barthel Index | 12 weeks
  To assess whether MR-001 improves activities of daily living in chronic stroke patients with gait deficit
PROMIS Social Isolation Scale | 12 weeks
  To assess whether MR-001 improves social isolation in patients with chronic stroke with gait deficit
Trail Making Tests A & B | 12 weeks
  To assess whether MR-001 improves cognition and executive in patients with chronic stroke with gait deficit

OTHER OUTCOMES:
6 Minute Walk Test (6MWT) | At 36 weeks
  To assess change in walking endurance of persons who are re-introduced to a second round of treatment with the intervention
Timed Up and Go (TUG) | 12 weeks
  To assess change in mobility after 12 weeks of intervention
Timed Up and Go (TUG) | At 36 weeks
  To assess change in mobility of persons who are re-introduced to a second round of treatment with the intervention
All-cause HCRU | Baseline to 52 weeks
  To assess change in all-cause healthcare resource utilization
All-cause hospitalizations and emergency department visits | Baseline to 52 weeks
  To assess change in all-cause hospitalizations and emergency department visits

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bethoux, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Curavit Clinical Research - DECENTRALIZED CLINICAL TRIAL, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor SR, Awad LN, Carlowicz CA, Maricich YA, Finklestein SP, Riley EH, Harris BA, Pohlig RT, Bethoux FA. Outcomes and Health Economics of Stroke using Rhythmic Auditory Stimulation (OrcHESTRAS): a protocol for a pragmatic, decentralized, longitudinal, multi-phase, withdrawal with randomized re-treatment trial of MR-001 in chronic stroke. Trials. 2026 Jan 8;27(1):108. doi: 10.1186/s13063-025-09415-3. PMID 41501870